CLINICAL TRIAL: NCT03881007
Title: A Double-blind Single Center, Crossover, Randomized Controlled Trial of Antibacterial vs. Placebo Mouthwash to Reduce the Incidence of Gonorrhea/Chlamydia/Syphilis in MSM Taking HIV Pre-exposure Prophylaxis (PrEP)
Brief Title: A Trial to Compare Antibacterial vs. Placebo Mouthwash to Reduce the Incidence of Sexually Transmitted Infections (STIs) in Men Who Have Sex With Men (MSM) Taking HIV Pre-Exposure Prophylaxis (PrEP)
Acronym: PReGo
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: An interim analysis, planned because of the influence of the COVID-lockdown, showed the LCM mouthwash did not affect the incidence of Ng, Ct and syphilis.
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: ITM201801
Record Dates: First submitted 2019-03-13; First posted 2019-03-19 (Actual); Results first posted 2021-04-06 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-04

CONDITIONS: Sexually Transmitted Diseases
Keywords: Gonorrhea; Syphilis; Chlamydia; Listerine; STI
MeSH Terms: conditions — Sexually Transmitted Diseases; Gonorrhea; Syphilis; Chlamydia Infections | interventions — Mouthwashes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LCM, then placebo (Experimental): Mouthwash with LCM for 3 months followed by mouthwash with placebo for 3 months.
  Interventions: Other: Mouthwash with LCM; Other: Mouthwash with placebo
- Placebo, then LCM (Experimental): Mouthwash with placebo for 3 months followed by mouthwash with LCM for 3 months
  Interventions: Other: Mouthwash with LCM; Other: Mouthwash with placebo

INTERVENTIONS:
Other: Mouthwash with LCM — Subjects will mouthwash daily with LCM and before/after sex
Other: Mouthwash with placebo — Subjects will mouthwash daily with placebo and before/after sex

SUMMARY:
The study involves a randomized placebo controlled trial that aims to assess if a mouthwash (Listerine cool mint, LCM) is able to reduce the cumulative incidence of gonorrhoea (Ng), chlamydia (Ct) and syphilis in men who have sex with men and receiving preexposure prophylaxis (PrEP) at the Institute of Tropical Medicine (ITM).

DETAILED DESCRIPTION:
The study aims to assess if there is a difference in the incidence rate of gonorrhea, chlamydia and syphilis detected at any site whilst individuals are on daily and pre/post sex Listerine cool mint (LCM) vs. placebo mouthwash.

The study has a double-blind, cross-over design, in which subjects will be screened at the ITM and, if eligible, will be enrolled and randomized to group 1 (LCM) or group 2 (placebo). After 3 months, a crossover will occur and subjects will switch to the other intervention. Each participant will therefore be enrolled for 6 months (2 x 3 months, no wash out period).

Subjects will be recruited from the existing PrEP cohort at the Institute of Tropical Medicine Antwerp. A total of 320 subjects will be recruited (160 in each arm).

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 or more
* Enrolled in Belgian PrEP program at ITM
* Has had sex with another man in the previous year
* Has had a symptomatic or asymptomatic STI (Ct/Ng/syphilis) in the previous 2 years
* Willing to be enrolled in the cohort for 6 months and attend 3 monthly follow up visits
* Willing to comply with the mouthwash study schema and willing to ask their casual partners to mouthwash pre- and post-sex
* Prepared to fill out the online diary once a week
* Able and willing to provide written informed consent

Exclusion Criteria:

* Currently using a mouthwash and unwilling to cease use of this mouthwash
* Enrolment in another interventional trial
* Tests HIV positive at screening

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 343 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Kenyon, MD, Principal Investigator — Institute of Tropical Medicine Antwerp
Locations (1):
- Institute of Tropical Medicine, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Data sharing for the PreGo trial will comply with ITMs Data Sharing Policy.
  Study data might be made available for secondary research and analyses to external researchers by means of a managed access procedure within 12 months of publication date. Because of privacy concerns, access requests will be reviewed and approved prior to release by ITMs Data Access Committee. Requests for access can be made centrally through:
  https://www.itg.be/E/data-sharing-open-access The possibility of sharing (anonymized) study data is also mentioned in the Informed Consent Form and approved by the Ethics Committees that approved the initial PreGo clinical trial protocol.
Supporting Information: Study Protocol, SAP
Time Frame: Available in clinicaltrials.gov

REFERENCES:
- [Derived] Akomoneh EA, Laumen JGE, Abdellati S, Van Dijck C, Vanbaelen T, Britto XB, Manoharan-Basil SS, Kenyon C. The Discovery of Oropharyngeal Microbiota with Inhibitory Activity against Pathogenic Neisseria gonorrhoeae and Neisseria meningitidis: An In Vitro Study of Clinical Isolates. Microorganisms. 2022 Dec 16;10(12):2497. doi: 10.3390/microorganisms10122497. PMID 36557750
- [Derived] Van Dijck C, Tsoumanis A, Rotsaert A, Vuylsteke B, Van den Bossche D, Paeleman E, De Baetselier I, Brosius I, Laumen J, Buyze J, Wouters K, Lynen L, Van Esbroeck M, Herssens N, Abdellati S, Declercq S, Reyniers T, Van Herrewege Y, Florence E, Kenyon C. Antibacterial mouthwash to prevent sexually transmitted infections in men who have sex with men taking HIV pre-exposure prophylaxis (PReGo): a randomised, placebo-controlled, crossover trial. Lancet Infect Dis. 2021 May;21(5):657-667. doi: 10.1016/S1473-3099(20)30778-7. Epub 2021 Mar 4. PMID 33676596

RESULTS

PARTICIPANT FLOW:
Groups:
- LCM (Intervention), Then Placebo: Mouthwash with Listerine Cool Mint: Subjects will mouthwash daily with LCM and before/after sex for 3 months and after 3 months they will switch to the placebo.
- Placebo, Then LCM (Intervention): Mouthwash with placebo: Subjects will mouthwash daily with placebo and before/after sex during 3 months and after 3 months they will switch to the LCM mouthwash.
Period: First 3 Months
Arm/Group | LCM (Intervention), Then Placebo | Placebo, Then LCM (Intervention)
Started | 172 | 171
Completed | 121 | 119
Not Completed | 51 | 52
Period: Last 3 Months
Arm/Group | LCM (Intervention), Then Placebo | Placebo, Then LCM (Intervention)
Started | 121 | 119
Completed | 77 | 74
Not Completed | 44 | 45

BASELINE CHARACTERISTICS:
Groups:
- LCM (Intervention), Then Placebo: Mouthwash with Listerine Cool Mint: Subjects will mouthwash daily with LCM and before/after sex for 3 months and then switch to placebo mouthwash for 3 months.
- Placebo, Then LCM: Mouthwash with placebo: Subjects will mouthwash daily with placebo and before/after sex for 3 months and then switch to LCM mouthwash for 3 months.
- Total: Total of all reporting groups
Arm/Group | LCM (Intervention), Then Placebo | Placebo, Then LCM | Total
Number analyzed (Participants) | 172 | 171 | 343
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 39 [31 to 48] | 40 [33.5 to 47] | 40 [32 to 47.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 172 | 171 | 343
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Sexually Transmitted Infection (STI) history (last 24 months) [Count of Participants; unit: Participants]
  Any STI | 172 | 171 | 343
  Chlamydia | 89 | 82 | 171
  Gonorrhea | 100 | 117 | 217
  Syphilis | 75 | 66 | 141
  Other | 15 | 21 | 36
Antibiotics use (last 6 months) [Count of Participants; unit: Participants]
  Any antibiotics | 140 | 136 | 276
  Macrolides | 71 | 86 | 157
  Beta-lactam | 111 | 121 | 232
  Fluoroquinolones | 4 | 3 | 7
  Tetracyclines | 47 | 30 | 77
  Other | 0 | 2 | 2
Number of main partners (last 3 months) [Median (Inter-Quartile Range); unit: Main partners] | 1 [0 to 2] | 1 [0 to 1] | 1 [0 to 1]
Number of casual partners (last 3 months) [Median (Inter-Quartile Range); unit: casual partners] | 10 [5 to 19] | 10 [5 to 20] | 10 [5 to 20]
Condom use with casual partners [Count of Participants; unit: Participants]
  0-24% | 50 | 62 | 112
  25-49% | 42 | 34 | 76
  50-74% | 31 | 26 | 57
  75-100% | 44 | 42 | 86

OUTCOME MEASURES:

1. Primary Outcome: Patient Counts of Ng Plus Ct Plus Syphilis in Each Study Arm for Each Period
Description: The sum of new diagnoses of Gonnorhea (Ng), Chlamydia (Ct) and syphilis in a 3 month period on LCM/placebo. Each participant can only contribute one diagnosis of Ct and one diagnosis of Ng per visit - regardless of number of sites infected. Thus each participant can contribute up to 3 diagnoses (Ct/Ng/syphilis) at each visit. The diagnosis of Ng and Ct will be made via molecular testing and syphilis via Rapid Plasma Reagin test (RPR) and Treponema Pallidum Antibodies tests (TPA) according to currently used European case definitions.
Time Frame: 3-month period following each intervention
Population: Intention-to-treat population. LCM (intervention) has a total of 195 participants (121 during the first 3 months and 74 during the last 3 months). The placebo arm had a total of 196 participants (119 during the first 3 months and 77 during the last 3 months).
Measure: Count of Participants; unit: Participants
Groups:
- LCM (Intervention): Mouthwash with Listerine Cool Mint: Subjects will mouthwash daily with LCM and before/after sex
- Placebo: Mouthwash with placebo: Subjects will mouthwash daily with placebo and before/after sex
Arm/Group | LCM (Intervention) | Placebo
Number analyzed (Participants) | 195 | 196
Participants
  First 3 months : Any STI: number analyzed (Participants) | 121 | 119
  First 3 months : Any STI | 36 | 33
  First 3 months : Chlamydia: number analyzed (Participants) | 121 | 119
  First 3 months : Chlamydia | 19 | 18
  First 3 months : Gonorrhea: number analyzed (Participants) | 121 | 119
  First 3 months : Gonorrhea | 19 | 17
  First 3 months : Syphilis: number analyzed (Participants) | 121 | 119
  First 3 months : Syphilis | 2 | 6
  Last 3 months : Any STI: number analyzed (Participants) | 74 | 77
  Last 3 months : Any STI | 27 | 21
  Last 3 months : Chlamydia: number analyzed (Participants) | 74 | 77
  Last 3 months : Chlamydia | 11 | 10
  Last 3 months : Gonorrhea: number analyzed (Participants) | 74 | 77
  Last 3 months : Gonorrhea | 14 | 8
  Last 3 months : Syphilis: number analyzed (Participants) | 74 | 77
  Last 3 months : Syphilis | 4 | 4
Statistical Analysis 1: Comparison: LCM (Intervention) vs Placebo; Test type: Superiority; p = 0.359, Mixed Models Analysis; Incidence rate ratio = 1.17, 95% CI 2-sided [0.84 to 1.64]

2. Secondary Outcome: Difference in Incidence Rate of Pharyngeal Ng Between Each Study Arm for Each Period
Description: Incidence rate of new pharyngeal Ng cases in each allocation arm for each study period of 3 months.
Time Frame: 3-month period following each intervention
Population: as for outcome 1
Measure: Number; unit: diagnoses
Arm/Group | LCM (Intervention) | Placebo
Number analyzed (Participants) | 195 | 196
diagnoses
  First 3 months: number analyzed (Participants) | 121 | 119
  First 3 months | 8 | 2
  Last 3 months: number analyzed (Participants) | 74 | 77
  Last 3 months | 3 | 0
Statistical Analysis 1: Comparison: LCM (Intervention) vs Placebo; Test type: Superiority; p = 0.024, Mixed Models Analysis; Incidence rate ratio = 5.78, 95% CI 2-sided [1.52 to 136.56]

3. Secondary Outcome: Difference in Incidence Rate of Ct (Combined Pharyngeal, Urethral and Rectal) Between Each Study Arm for Each Period
Description: Incidence rate of new Ct cases in each allocation arm (LCM and placebo) for each study period of 3 months.
Time Frame: 3-month period following each intervention
Population: as for outcome 1
Measure: Number; unit: diagnoses
Arm/Group | LCM (Intervention) | Placebo
Number analyzed (Participants) | 195 | 196
diagnoses
  First 3 months: number analyzed (Participants) | 121 | 119
  First 3 months | 19 | 18
  Last 3 months: number analyzed (Participants) | 74 | 77
  Last 3 months | 11 | 10
Statistical Analysis 1: Comparison: LCM (Intervention) vs Placebo; Test type: Superiority; p = 0.774, Mixed Models Analysis; Incidence rate ratio = 1.09, 95% CI 2-sided [0.61 to 1.95]

4. Secondary Outcome: Difference in Incidence Rate of Syphilis Between Periods on LCM vs. Placebo
Description: Incidence rate of new syphilis cases in each allocation arm (LCM and placebo) for each study period of 3 months.
Time Frame: 3-month period following each intervention
Population: as for outcome 1
Measure: Number; unit: diagnoses
Arm/Group | LCM (Intervention) | Placebo
Number analyzed (Participants) | 195 | 196
diagnoses
  First 3 months: number analyzed (Participants) | 121 | 119
  First 3 months | 2 | 6
  Last 3 months: number analyzed (Participants) | 74 | 77
  Last 3 months | 4 | 4
Statistical Analysis 1: Comparison: LCM (Intervention) vs Placebo; Test type: Superiority; p = 0.323, Mixed Models Analysis; incidence rate ratio = 0.59, 95% CI 2-sided [0.2 to 1.63]

5. Secondary Outcome: Proportion of Days That Mouthwash is Used on a Daily Basis and Proportion of Casual Sex Contacts When Mouthwash is Used Pre or Post Sex
Description: Daily: Proportion of days in study used mouthwash at least daily Post sex: Proportion of casual sexual contacts in study when mouthwash used post sex.
  Pre sex: proportion of casual sexual contacts in study when mouthwash used pre sex
Time Frame: 6-month period
Population: Intention-to-treat population.LCM (intervention) has a total of 195 participants (121 during the first 3 months and 74 during the last 3 months). The placebo arm had a total of 196 participants (119 during the first 3 months and 77 during the last 3 months).
Measure: Count of Participants; unit: Participants
Arm/Group | LCM (Intervention) | Placebo
Number analyzed (Participants) | 195 | 196
Participants
  Month 3 daily use: number analyzed (Participants) | 121 | 119
  Month 3 daily use: 0-24% | 11 | 14
  Month 3 daily use: 25-49% | 8 | 9
  Month 3 daily use: 50-74% | 17 | 14
  Month 3 daily use: 75-100% | 80 | 79
  Month 3 daily use: Missing | 5 | 3
  Month 6 daily use: number analyzed (Participants) | 74 | 77
  Month 6 daily use: 0-24% | 6 | 6
  Month 6 daily use: 25-49% | 4 | 5
  Month 6 daily use: 50-74% | 9 | 11
  Month 6 daily use: 75-100% | 15 | 9
  Month 6 daily use: Missing | 40 | 46
  Month 3 pre-sex: number analyzed (Participants) | 121 | 119
  Month 3 pre-sex: 0-24% | 30 | 36
  Month 3 pre-sex: 25-49% | 15 | 18
  Month 3 pre-sex: 50-74% | 20 | 19
  Month 3 pre-sex: 75-100% | 49 | 41
  Month 3 pre-sex: Missing | 7 | 5
  Month 6 pre-sex: number analyzed (Participants) | 74 | 77
  Month 6 pre-sex: 0-24% | 19 | 13
  Month 6 pre-sex: 25-49% | 13 | 15
  Month 6 pre-sex: 50-74% | 13 | 18
  Month 6 pre-sex: 75-100% | 25 | 24
  Month 6 pre-sex: Missing | 4 | 7
  Month 3 post-sex: number analyzed (Participants) | 121 | 119
  Month 3 post-sex: 0-24% | 31 | 38
  Month 3 post-sex: 25-49% | 16 | 16
  Month 3 post-sex: 50-74% | 22 | 26
  Month 3 post-sex: 75-100% | 45 | 34
  Month 3 post-sex: Missing | 7 | 5
  Month 6 post-sex: number analyzed (Participants) | 74 | 77
  Month 6 post-sex: 0-24% | 22 | 14
  Month 6 post-sex: 25-49% | 13 | 17
  Month 6 post-sex: 50-74% | 14 | 18
  Month 6 post-sex: 75-100% | 21 | 21
  Month 6 post-sex: Missing | 4 | 7

6. Secondary Outcome: Difference in Incidence Rate of Ng Plus Ct Plus Syphilis Between LCM and Placebo After Controlling for Adherence With Daily and Pre/Post Sex Mouthwash
Description: Incidence rate of Ng, Ct and syphilis between both groups (LCM and placebo) post controlling for adherence to mouthwash
Time Frame: 3-month period following each intervention
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | LCM (Intervention) | Placebo
Number analyzed (Participants) | 195 | 196
Participants
  First 3 months: Any STIs: number analyzed (Participants) | 121 | 119
  First 3 months: Any STIs | 36 | 33
  First 3 months: Chlamydia: number analyzed (Participants) | 121 | 119
  First 3 months: Chlamydia | 19 | 18
  First 3 months: Gonorrhea: number analyzed (Participants) | 121 | 119
  First 3 months: Gonorrhea | 19 | 17
  First 3 months: Syphilis: number analyzed (Participants) | 121 | 119
  First 3 months: Syphilis | 2 | 6
  Last 3 months: Any STI: number analyzed (Participants) | 74 | 77
  Last 3 months: Any STI | 27 | 21
  Last 3 months: Chlamydia: number analyzed (Participants) | 74 | 77
  Last 3 months: Chlamydia | 11 | 10
  Last 3 months: Gonorrhea: number analyzed (Participants) | 74 | 77
  Last 3 months: Gonorrhea | 14 | 8
  Last 3 months: Syphilis: number analyzed (Participants) | 74 | 77
  Last 3 months: Syphilis | 4 | 4
Statistical Analysis 1: Comparison: LCM (Intervention) vs Placebo; Test type: Superiority; p = 0.279, Mixed Models Analysis; Incidence rate ratio = 1.21, 95% CI 2-sided [0.86 to 1.72]

7. Secondary Outcome: Difference in Cumulative Numbers of Antibiotics Used Between Periods on LCM vs. Placebo
Description: Cumulative number of antibiotics used between both groups (LCM and placebo) for each period
Time Frame: 3-month period following each intervention
Population: The overall number of participants analyzed is for both study periods. The number analyzed per row is the number of participants analyzed per period. LCM (intervention) has a total of 195 participants (121 during the first 3 months and 74 during the last 3 months). The placebo arm had a total of 196 participants (119 during the first 3 months and 77 during the last 3 months).
Measure: Count of Participants; unit: Participants
Arm/Group | LCM (Intervention) | Placebo
Number analyzed (Participants) | 195 | 196
Participants
  Month 3: number analyzed (Participants) | 121 | 119
  Month 3 | 49 | 55
  Month 6: number analyzed (Participants) | 74 | 77
  Month 6 | 39 | 35

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were collected over the whole study duration (6 months)
Description: Adverse events are reported per intervention. LCM (intervention) has a total of 195 participants (121 during the first 3 months and 74 during the last 3 months). The placebo arm had a total of 196 participants (119 during the first 3 months and 77 during the last 3 months).
Groups:
- LCM (Intervention): Mouthwash with Listerine Cool Mint: Subjects will mouthwash daily with LCM and before/after sex. The total of participants at risk for the LCM intervention is 195 (121 in first 3 months and 77 in last 3 months).
- Placebo: Mouthwash with placebo: Subjects will mouthwash daily with placebo and before/after sex. The total of participants at risk for the LCM intervention is 196 (119 in first 3 months and 74 in last 3 months).
Arm/Group | LCM (Intervention) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/195 | 0/196
Serious Adverse Events (participants affected / at risk) | 1/195 | 3/196
Other Adverse Events (participants affected / at risk) | 45/195 | 30/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LCM (Intervention) (N=195) | Placebo (N=196)
Ludwig Angina (Infections and infestations) | 1 (1) | 0 (0)
Suicidal depression (Psychiatric disorders) | 0 (0) | 1 (1)
Testis carcinoma (Reproductive system and breast disorders) | 0 (0) | 1 (1)
HIV (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LCM (Intervention) (N=195) | Placebo (N=196)
Dental caries (Gastrointestinal disorders) | 19 (19) | 12 (12)
Tooth discoloration (Gastrointestinal disorders) | 26 (26) | 18 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-01-08): https://cdn.clinicaltrials.gov/large-docs/07/NCT03881007/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/07/NCT03881007/SAP_001.pdf